CLINICAL TRIAL: NCT05657912
Title: A Continuous ECG Monitoring Data Collection Study in Patients Undergoing Transcatheter Aortic Valve Replacement (TAVR) to Evaluate the Performance of the Cara Monitor Conduction Disturbance Risk Score (CDRS).
Brief Title: Cara CDRS (Conduction Disturbance Risk Score) 1.0
Acronym: CDRS
Status: Completed | Type: Observational
Sponsor: Cara Medical Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Cara 1.0
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-02

CONDITIONS: Transcatheter Aortic Valve Replacement
MeSH Terms: interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- ECG Monitoring -TAVR patients: Continuous ECG monitoring of Conduction Disturbances in patients undergoing TAVR procedure
  Interventions: Device: ECG monitoring

INTERVENTIONS:
Device: ECG monitoring — Continuous ECG monitoring of Conduction Disturbances in patients undergoing TAVR procedure

SUMMARY:
Prospective, non-randomized, multicenter data collection study. Eligible TAVR patients will be enrolled in the study.

Cardiac conduction disturbances (CD) requiring permanent pacemaker implantation (PPM) or causing new-onset CD are frequent complications of TAVR that have been shown to be associated with increased mortality and re-hospitalization rates.

The purpose of the study is to collect continuous ECG data in order to validate the performance of the Cara Conduction Disturbance Risk Score (CDRS) in patients undergoing transcatheter aortic valve replacement (TAVR).

Subjects will be studied during the TAVR procedure and their ECG recordings according to the study schedule below of pre-, during, and after the TAVR procedure up to 14/30 days FU will be collected.

600 patients will be enrolled in this study with the hypothesis that Cara can deliver a statistically significant conduction disturbance risk stratification for patients undergoing TAVR.

No investigation intervention is planned during this study. The Cara System analysis will be performed offline.

DETAILED DESCRIPTION:
TAVR will be performed using site investigators' best practices including the use of standard-of-care catheters, devices, imaging, and monitoring modalities.

Data will be collected to include the following patients' measures during this study:

1. Pre-procedure

   1. Demographics
   2. Medical history
   3. Cardiac CT
   4. 12 lead ECG
2. Procedure

   1. Continuous 3-12 lead Holter will be supplied, data will be collected and analyzed by the study sponsor
   2. Fluoroscopy (captured automatically by video system )
   3. Device manufacturer (type) and size
3. Post-procedure (in hospital)

   a. Continuous 1-3 lead Holter for 14 days will be supplied, and the data from the Holter recordings will be collected from the patient's home and analyzed.
4. Post-procedure (discharge)

   a. 12 lead ECG
5. Patients will be followed according to the current medical practice.

Data to be collected during the FU :

a. 12 lead ECG at 14/30 days

The data collected from the study will be used to evaluate the performance Cara System, a conduction disturbance monitor that provides an indication of conduction disturbances during TAVR procedures.

Conduction Disturbances (CD) outcome will be subdivided into:

1. PPM or High-Grade AV Block (HGAVB)
2. All other new onsets (or deterioration) of CD that are not listed in #1
3. No new onset CD

ELIGIBILITY:
Inclusion Criteria:

* Must meet be ≥ 18 years of age.
* Must meet indications for TAVR using approved devices
* Provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
* Willing to comply with specified follow-up evaluations.
* Must meet the legal minimum age to provide Informed Consent based on local regulatory requirements.

Exclusion Criteria:

* Any implanted device or an indication for treatment with a rhythm management device (i.e., pacemaker, Cardiac Resynchronization Therapy (CRT), or Cardiac Resynchronization Therapy with cardioverter-defibrillator (CRT-D) at baseline.
* Any contraindication to the TAVR procedure according to the instructions for use.
* Less than the legal age of consent, legally incompetent, or otherwise vulnerable.
* Planned treatment with any other investigational device, drug, or procedure (excluding registries) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 patients undergoing TAVR will be enrolled at the investigational sites.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Estimated reduction of New Onset Conduction Disturbances NOCD (percentage) at 14 days post TAVR while using Cara Monitor | 14 days
  Continuous ECG data collected during the TAVR procedure will be used to retrospectively evaluate the performance of the Cara monitor Conduction Disturbance Risk Score (CDRS) in patients post- TAVR procedure.
  Measured output:
  1. Patients who receive PaceMaker (PPM) 14 days following TAVr (PPM+)
  2. Patients that do not receive PaceMaker (PPM) 14 days following TAVr (PPM-)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Grinberg-Rashi, PhD, Study Chair — helenag@k2-medicalltd.com
Locations (3):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval, Québec, Canada
- Policlinico San Donato, Milan, Italy
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No